CLINICAL TRIAL: NCT05095116
Title: APT-1011 (Fluticasone ODT) Expanded Access Protocol for Patients With Eosinophilic Esophagitis
Brief Title: Expanded Access Protocol for Patients With Eosinophilic Esophagitis
Status: No longer available | Type: Expanded Access
Sponsor: Ellodi Pharmaceuticals, LP (Industry)
Responsible Party: Sponsor
Other Study IDs: SP-1011-004
Record Dates: First submitted 2021-10-14; First posted 2021-10-27 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Eosinophilic Esophagitis
Keywords: APT-1011; Esophagitis; Eosinophilic Esophagitis; Esophageal Diseases; Gastrointestinal Diseases; Gastroenteritis; Eosinophilia; Leukocyte Disorders; Hematologic Diseases; Hypersensitivity, Immediate; Hypersensitivity; Immune System Diseases; Fluticasone; Anti-Inflammatory Agents; Bronchodilator Agents; Autonomic Agents; Peripheral Nervous System Agents; Anti-Asthmatic Agents; Respiratory System Agents; Anti-Allergic Agents
MeSH Terms: conditions — Eosinophilic Esophagitis; Esophagitis; Esophageal Diseases; Gastrointestinal Diseases; Gastroenteritis; Eosinophilia; Leukocyte Disorders; Hematologic Diseases; Hypersensitivity, Immediate; Hypersensitivity; Immune System Diseases | interventions — APT-1011; Fluticasone

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: APT-1011 3 mg HS — APT-1011 is an orally disintegrating tablet that includes fluticasone propionate as its active ingredient.
  Other Names: fluticasone propionate

SUMMARY:
This expanded access program is an open-label, single-arm design where consenting patients may participate up until APT-1011 is commercially available in the relevant regions or the protocol is terminated by the Sponsor.

DETAILED DESCRIPTION:
Patients will receive a 120-day supply of APT-1011 and will attend scheduled clinic visits every 4 months. Telephone visits will be performed as needed. At each clinic visit (or additional telephone visit), adverse events (AEs) and concomitant medications will be collected. The Global EoE score will be collected at clinic visits.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥12 years of age at the time of informed consent
2. Signed ICF and willing and able to adhere to all procedures; signed assent form and parent/guardian ICF must also be collected for adolescents
3. Confirmed medical history of EoE
4. Adult and adolescent patients who are unable or ineligible to enroll in an APT-1011 clinical study or have failed available treatment options
5. Willing and able to adhere to the treatment regimen and visit schedule

Exclusion Criteria:

1. Have known contraindication, hypersensitivity, or intolerance to corticosteroids
2. Have signs and symptoms of adrenal suppression or hypercorticism
3. Use of potent CYP3A4 inhibitors (e.g., ritonavir and ketoconazole) are prohibited
4. Have current alcohol or drug abuse in the opinion of the Investigator
5. Female patients who are pregnant, breastfeeding, or planning to become pregnant while participating in the program
6. Female patients of child-bearing potential who are unable to comply with adequate contraception use during the program

Min Age: 12 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (35):
- United States (35):
  - Del Sol Research Management LLC, Tucson, Arizona
  - Arkansas Gastroenterology, North Little Rock, Arkansas
  - Ventura County Gastroenterology Medical Group Camarillo, Camarillo, California
  - FOMAT Medical Research, Glendale, California
  - United Medical Doctors, Murrieta, California
  - Medical Associates Research Group, San Diego, California
  - Peak Gastroenterology Associates, Colorado Springs, Colorado
  - Western States Clinical Research Inc, Wheat Ridge, Colorado
  - Nuvance Health Medical Practice Ct, Inc., Danbury, Connecticut
  - Medical Research Center of Connecticut, Hamden, Connecticut
  - Nature Coast Clinical Research, Inverness, Florida
  - Endoscopic Research, Inc., Orlando, Florida
  - Summit Clinical Research, Athens, Georgia
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - MGG Group Co., Inc., Chevy Chase, Maryland
  - Gastro Center of Maryland, Columbia, Maryland
  - Boston Specialists, Boston, Massachusetts
  - Clinical Research Institute of Michigan LLC, Chesterfield, Michigan
  - Henry Ford Health System, Novi, Michigan
  - West Michigan Clinical Research Center, Wyoming, Michigan
  - MNGI Digestive Health, P.A., Minneapolis, Minnesota
  - Minnesota Gastroenterology PA Plymouth Endoscopy Center Clinic, Plymouth, Minnesota
  - Clinical Research Professionals, Chesterfield, Missouri
  - Bozeman Health Clinical Research, Bozeman, Montana
  - Clinical and Translational Research Center (CTRC), Chapel Hill, North Carolina
  - Carolina Research, Greenville, North Carolina
  - Gastro Health Research, Cincinnati, Ohio
  - Bernstein Clinical Research Center, LLC, Cincinnati, Ohio
  - Great Lakes Gastroenterology, Mentor, Ohio
  - Northshore Gastroenterology Research LLC, Westlake, Ohio
  - Vital Prospects Clinical Research Institute, P.C., Tulsa, Oklahoma
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Regional Gastroenterology Associates of Lancaster, Ltd., Wyomissing, Pennsylvania
  - Rapid City Medical Center LLP, Rapid City, South Dakota
  - GI Alliance, Garland, Texas